CLINICAL TRIAL: NCT01173783
Title: Deutsches Device Qualitätsregister
Status: Completed | Type: Observational
Sponsor: Stiftung Institut fuer Herzinfarktforschung (Other)
Responsible Party: Sponsor
Other Study IDs: DEVICE
Record Dates: First submitted 2010-07-29; First posted 2010-08-02 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-06

CONDITIONS: Heart Failure
Keywords: Heart failure; Cardiac insufficiency; Implantable Cardioverter/Defibrillator; Cardiac Resynchronization therapy; ICD; CRT; Register
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
It is the aim of this register to document the development of therapies by implantation of Cardioverter/Defibrillators (ICDs) and/or Cardiac Resynchronization therapy (CRT)-Systems.

DETAILED DESCRIPTION:
The possibility of evaluation of successes as well as of the complications of these therapies is needed to make quality management possible. Every German Center, implanting ICDs or CRT-devices, is encouraged to contribute to this register; data are collected by use of an electronical CRF.

ELIGIBILITY:
Inclusion Criteria:

* The Device register will include all consecutive patients with an intended implantation of an ICD / CRT.

Exclusion Criteria:

* Missing signed informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all consecutive patients with an intended implantation of an ICD / CRT.
Sampling Method: Non-Probability Sample
Enrollment: 4008 (Actual)
Dates: Start 2007-03; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Characterize consecutive patients with initial implantation of ICD or CRT in hospital daily routine in Germany | 01/03/2007-12/31/2011

SECONDARY OUTCOMES:
Specification of the device and the realization of the implantation as well as the success of the operation | 01/03/2007-12/31/2011
Documentation of further interventions needed after the Index Event during hospital stay | 01/03/2007-12/31/2011
Documentation of hospital mortality and non-fatal complications | 01/03/2007-12/31/2011
Documentation of the 1-year mortality and non-fatal complications | 01/03/2007-12/31/2011
Documentation of the dispensary of shocks within one year | 01/03/2007-12/31/2011
Documentation of symptomatology and number of hospitalizations | 01/03/2007-12/31/2011
Documentation of medication therapy after 12 months | 01/03/2007-12/31/2011

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Senges, MD, Principal Investigator — Stiftung Institut fuer Herzinfarktforschung
Locations (7):
- Germany (7):
  - Vivantes Klinikum Am Urban, Berlin
  - Städtische Kliniken Bielefeld, Bielefeld
  - St. Marien Hospital, Bonn
  - Evangelisches Krankenhaus Düsseldorf, Düsseldorf
  - Asklepios Klinik St Georg, Hamburg
  - St. Vincentius Klinikan AG, Karlsruhe
  - Klinikum Villingen-Schwenningen, Villingen-Schwenningen

IPD SHARING:
Plan to Share IPD: No